CLINICAL TRIAL: NCT05393960
Title: Effects of Lumbosacral Mobility Program on Muscle Length in Sedentary Young Adults With Tight Hamstrings
Brief Title: Effects of Lumbosacral Mobility Program on Tight Hamstrings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/ 22/0138 Kanwal
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Hamstring Tightness
Keywords: manual therapy; lumbar mobility; mobilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization (Experimental): Lumbosacral manual therapy mobilization
  Interventions: Other: Lumbosacral manual therapy mobilization, lumber mobility exercises and home based self strechings program.
- Stretching program (Other): home based self strechings program
  Interventions: Other: home based self strechings program only.

INTERVENTIONS:
Other: Lumbosacral manual therapy mobilization, lumber mobility exercises and home based self strechings program. — Manual therapy, mobility exercise therapy and a home-based self-stretching program. Manual mobilization postero-anterior glides at lumber facets joints, Transverse glides at spinous process & Posterior-anterior glides at SI joint. Glides will be performed 3 times with 5 repetitions. Mobility exercise therapy.
  Arms: Mobilization
Other: home based self strechings program only. — Home based self-stretching program includes 3 repetitions of 15 seconds duration stretch (with 20 seconds rest between each repetition). Repeat stretching exercises twice a day for 3 alternate days for 1 week. Piriformis stretch: in supine crook lying, placing the lateral side of the foot over the contralateral knee and pulling towards the chest with the hands. Quadriceps stretch: stand on your left leg, one knee touching the other, hold a chair or the wall to keep you steady if needed, grab your right foot, using your right hand, and pull it towards your butt. Hamstring stretch: To stretch the right leg, sit on the ground with the left leg bent at the knee with the foot facing inward. This is called the butterfly position. Extend the right leg, keeping it slightly bent at the knee. Bend forward at the waist, making sure to keep the back straight.
  Arms: Stretching program

SUMMARY:
The study will be randomized controlled trial to determine the effects of lumbosacral mobility program on muscle length in sedentary young adults with tight hamstrings. Only the eligible subjects who fulfill the inclusion criteria will be included in the study. A sample of 78 subjects will be taken and randomly allocated into two groups with 39 each. Group A will be given three treatments. Manual therapy, mobility exercise therapy and home based self stretching program. Manual therapy mobilization posterior-anterior glides at lumber facets joints, transverse glides at spinous process & Posterior-anterior glides at SI joint. Glides will be performed 3 times with 5 repetitions. Mobility exercise therapy (Single knee to chest, double knee to chest, Lumbar rotation, Lumbar extension, Pelvic tilting). A total of 30 min sessions three times a week on alternate days for 1 week & home-based self-stretches program twice a day for three times a week on alternate days for 1 week. Group B will be given home-based self-stretching program twice a day for three times a week on alternate days for 1 week .The baseline values of all the dependent variable will be recorded on day one and at the end of the 1-week treatment session, using goniometry, active and passive knee extension test, passive straight leg raising and lower extremity functional scale will be used

DETAILED DESCRIPTION:
The hamstring muscle group consists of four muscles (semitendinosus, semimembranosus, biceps femoris long head, biceps femoris short head). It's a two-joint muscle working simultaneously to act as a hip extensor and knee flexor. It also functions to maintain the stability of the knee joint. The hamstring plays important role in daily activities like running & walking. A lot of factors affecting hamstring function, one of them is flexibility, it is defined as the extent to which muscle length contributes to maximal joint range of motion. It is a well-known muscle of has a shortening tendency. There are many methods for treating hamstrings flexibility/tightness/shortening. Routinely, physiotherapists are using stretching & strengthening exercises, instruments assisted in soft tissue mobilization. The current study focuses on two treatments manual therapy & lumber mobility exercises

ELIGIBILITY:
Inclusion Criteria:

* Age 20-30 years
* Sedentary life style
* BMI < 23 non-obese
* Hamstring shortness ≥ 20° using the active knee extension test (aket)
* No history of orthopedic/neurologic disorders in the lower extremity
* No history of back pain in last 2 weeks
* No contraindication for using manual therapy
* No joint limitation in the lower extremities

Exclusion Criteria:

* Any systemic soft tissue and bony disease
* Fracture
* Neuropathy
* Congenital deformities of spine

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Active knee extension test | 1 Week
  A reliable tool for hamstring length measurement. Subject is in supine lying position on examination table while other leg is in extension position stabilized with two strap. One across midthigh and other across pelvis ( to prevent compensatory movements ) subject were asked to extens the knee until stretch sensation felt ayt posterior aspect of thigh. Note the range with goniometer
Passive knee extension test | 1 Week
  A reliable tool for hamstring length measurement. Subject is in supine lying position on examination table while other leg is in extension position stabilized with two strap. One across midthigh and other across pelvis ( to prevent compensatory movements ) now passively extend subject's knee until stretch sensation felt at posterior aspect of thigh. Note the range with goniometer.
Goniometry | 1 Week
  It is an affordable & available tool for measurement of joint range of motion in degrees. (18) Passive Straight Leg Raise (SLR) test Subject is asked to maintain a position of supine lying on examination bed. Then passive SLR is performed by lifting subject heel. ( knee remains in extension ) pelvis should remain stabilize. look for the point at which discomfort starts. Note the range.
LEFS | 1 Week
  It is well known validated tool used to assess the functioning of lower extremity. It's a 20 question test which further subgroups into 4. Questions based on physical activity of lower extremity

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- FMH Institute of allied health sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stepien K, Smigielski R, Mouton C, Ciszek B, Engelhardt M, Seil R. Anatomy of proximal attachment, course, and innervation of hamstring muscles: a pictorial essay. Knee Surg Sports Traumatol Arthrosc. 2019 Mar;27(3):673-684. doi: 10.1007/s00167-018-5265-z. Epub 2018 Oct 29. PMID 30374579
- [Background] Kellis E. Intra- and Inter-Muscular Variations in Hamstring Architecture and Mechanics and Their Implications for Injury: A Narrative Review. Sports Med. 2018 Oct;48(10):2271-2283. doi: 10.1007/s40279-018-0975-4. PMID 30117053
- [Background] Chang JS, Kayani B, Plastow R, Singh S, Magan A, Haddad FS. Management of hamstring injuries: current concepts review. Bone Joint J. 2020 Oct;102-B(10):1281-1288. doi: 10.1302/0301-620X.102B10.BJJ-2020-1210.R1. PMID 32993323
- [Background] Guruhan S, Kafa N, Ecemis ZB, Guzel NA. Muscle Activation Differences During Eccentric Hamstring Exercises. Sports Health. 2021 Mar;13(2):181-186. doi: 10.1177/1941738120938649. Epub 2020 Aug 28. PMID 32857686
- [Background] Medeiros DM, Cini A, Sbruzzi G, Lima CS. Influence of static stretching on hamstring flexibility in healthy young adults: Systematic review and meta-analysis. Physiother Theory Pract. 2016 Aug;32(6):438-445. doi: 10.1080/09593985.2016.1204401. Epub 2016 Jul 26. PMID 27458757
- [Background] Shamsi M, Mirzaei M, Shahsavari S, Safari A, Saeb M. Modeling the effect of static stretching and strengthening exercise in lengthened position on balance in low back pain subject with shortened hamstring: a randomized controlled clinical trial. BMC Musculoskelet Disord. 2020 Dec 4;21(1):809. doi: 10.1186/s12891-020-03823-z. PMID 33276764
- [Background] Osailan A, Jamaan A, Talha K, Alhndi M. Instrument assisted soft tissue mobilization (IASTM) versus stretching: A comparison in effectiveness on hip active range of motion, muscle torque and power in people with hamstring tightness. J Bodyw Mov Ther. 2021 Jul;27:200-206. doi: 10.1016/j.jbmt.2021.03.001. Epub 2021 Mar 11. PMID 34391234
- [Background] Gunn LJ, Stewart JC, Morgan B, Metts ST, Magnuson JM, Iglowski NJ, Fritz SL, Arnot C. Instrument-assisted soft tissue mobilization and proprioceptive neuromuscular facilitation techniques improve hamstring flexibility better than static stretching alone: a randomized clinical trial. J Man Manip Ther. 2019 Feb;27(1):15-23. doi: 10.1080/10669817.2018.1475693. Epub 2018 Aug 1. PMID 30692839
- [Background] Moon JH, Jung JH, Won YS, Cho HY. Immediate effects of Graston Technique on hamstring muscle extensibility and pain intensity in patients with nonspecific low back pain. J Phys Ther Sci. 2017 Feb;29(2):224-227. doi: 10.1589/jpts.29.224. Epub 2017 Feb 24. PMID 28265144
- [Background] Sadler SG, Spink MJ, Ho A, De Jonge XJ, Chuter VH. Restriction in lateral bending range of motion, lumbar lordosis, and hamstring flexibility predicts the development of low back pain: a systematic review of prospective cohort studies. BMC Musculoskelet Disord. 2017 May 5;18(1):179. doi: 10.1186/s12891-017-1534-0. PMID 28476110